CLINICAL TRIAL: NCT02884271
Title: Intraoperative Cardiac Arrest: Incidence and Outcome
Brief Title: Cardiopulmonary Resuscitation in Operating Room
Acronym: CPR
Status: Recruiting | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Staff anesthesiologists in Department of Anaesthesiology and Intensive Care in Dokuz Eylul Universty Hospital, Dokuz Eylul University
Other Study IDs: 2482-GOA
Record Dates: First submitted 2016-08-17; First posted 2016-08-30 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Intraoperative Cardiac Arrest
Keywords: CPR; cardiac arrest; operating room
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cardiac arrest group: patients who develop intraoperative cardiac arrest
  Interventions: Procedure: cardiopulmonary resuscitation
- without cardiac arrest group: patients who don't develop intraoperative cardiac arrest

INTERVENTIONS:
Procedure: cardiopulmonary resuscitation — start cardiopulmonary resuscitation
  Groups: cardiac arrest group

SUMMARY:
In the last ten years patient safety during routine surgical interventions has increased; however as there is an increase in the number of specialized surgical interventions and high risk patients like elderly and emergency patients, the incidence of perioperative cardiac arrest has not reduced but remains fixed. The incidence of perioperative cardiac arrest varies from 4.3-34.6 for each 10,000 procedures. However as in a lot of other countries exact data are lacking also for Turkey. With this study the investigators want to start collecting data about intraoperative cardiac arrest in Turkey, starting at their institution The aim is to evaluate the incidence and outcome in the study. Secondary aim is to assess the causes of cardiac arrest in the operating room.

DETAILED DESCRIPTION:
Patient information will be collected on a form entitled "Data collection form" including all medications and interventions during cardiopulmonary resuscitation and routine daily used anesthesia registration form.

ELIGIBILITY:
Inclusion Criteria:

* All patients who develop cardiac arrest in the operating room

Exclusion Criteria:

* Absence of informed consent
* Patients arriving into the operating room with ongoing CPR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all patients who develop cardiac arrest in the operating room (including preoperative waiting area and postoperative recovery unit) Dokuz Eylul University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
incidence of intraoperative cardiac arrest | baseline
neurologic outcome of patients according to Cerebral performance category scale | until six months after return of spontaneous circulation

SECONDARY OUTCOMES:
causes of intraoperative cardiac arrest among participants/patients | baseline
  Probable causes of intraoperative cardiac arrest among participants/patients
  1. Trauma
  2. End stage liver disease and complications associated with liver transplantation
  3. Unable to wean from cardiopulmonary bypass
  4. Complications associated with cardiac surgery
  5. Ruptured aneurysm; abdominal or thoracic
  6. Technical complications: surgical and special procedures, central venous access
  7. Complications associated with automatic implantable cardiac defibrillator placement
  8. Hemorrhage
  9. Complications associated with radical cancer surgery
  10. Sepsis and multiple organ failure
  11. Perioperative myocardial infarction
  12. Complications associated with congenital heart defect
  13. Complications associated with neurosurgery
  14. Complications associated with Anaesthesia (anaphylaxis, difficult airway management/difficult ventilation, adverse drug, total spinal anaesthesia/bloc etc)

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Kuvaki, Professor, Principal Investigator — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes